CLINICAL TRIAL: NCT01313871
Title: Cross-sectional Study of Disease Severity and Treatment Patterns of Rheumatoid Arthritis, in Eastern Europe Middle East and North Africa
Brief Title: Assessment of the Disease Severity and Treatment Patterns of Rheumatoid Arthritis in Eastern Europe, Middle East and North African Countries (P08167)
Status: Withdrawn | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P08167
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants: Adults with a confirmed diagnosis of rheumatoid arthritis

SUMMARY:
The study will assess the disease severity and treatment patterns of rheumatoid arthritis in Eastern European, Middle Eastern, and North African countries.

ELIGIBILITY:
Inclusion Criteria :

* Confirmed diagnosis of rheumatoid arthritis, preferably based upon criteria established by the American College of Rheumatology (ACR) 1987
* clinical signs & symptoms
* data obtained from previous laboratory and instrumental examination, which may include but is not limited to: Radiography, Blood tests
* Written informed consent, signed before participation in the study.

Exclusion Criteria :

* Refusal to participate in the study
* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a confirmed diagnosis of rheumatoid arthritis
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with low, moderate, or high disease activity as assessed by the Disease Activity Score using 28 joint counts (DAS28) | Day of enrollment (Day 0)

SECONDARY OUTCOMES:
The number of participants with rheumatoid arthritis visiting participating sites in the course of one year | One year
Number of participants with different degrees of disability as assessed by the Health Assessment Questionnaire (HAQ). | Day of enrollment (Day 0)
Number of participants treated with non-steroidal anti-inflammatory drugs (NSAIDs), disease-modifying anti-rheumatic drugs (DMARDS), corticosteroids, and/or biologics | Day of enrollment (Day 0)